CLINICAL TRIAL: NCT03800134
Title: A Phase III, Double-blind, Placebo-controlled, Multi-center International Study of Neoadjuvant/Adjuvant Durvalumab for the Treatment of Patients With Resectable Stages II and III Non-small Cell Lung Cancer (AEGEAN)
Brief Title: A Study of Neoadjuvant/Adjuvant Durvalumab for the Treatment of Patients With Resectable Non-small Cell Lung Cancer
Acronym: AEGEAN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9106C00001; 2018-002997-29 (EudraCT Number)
Record Dates: First submitted 2018-12-07; First posted 2019-01-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Resectable Non-small Cell Lung Cancer, NSCLC, Carcinoma, Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — durvalumab; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel; Gemcitabine; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Durvalumab with platinum-based chemotherapy (Experimental): Patients will receive durvalumab 1500 mg in combination with platinum-based chemotherapy every 3 weeks for up to 4 cycles prior to surgery, followed by durvalumab 1500 mg monotherapy every 4 weeks for up to 12 cycles after surgery unless disease is deemed unresectable, disease recurrence, or unacceptable toxicity
  The platinum-based chemotherapy will be based on tumour histology and Investigator discretion:
  * cisplatin with pemetrexed
  * carboplatin with pemetrexed
  * carboplatin with paclitaxel
  * cisplatin with gemcitabine (or carboplatin with gemcitabine for patients who have comorbidities or who are unable to tolerate cisplatin per the investigator's judgment)
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Gemcitabine; Procedure: Surgery
- Arm 2: Placebo with platinum-based chemotherapy (Placebo Comparator): Patients will receive placebo in combination with platinum-based chemotherapy every 3 weeks for up to 4 cycles prior to surgery, followed by placebo monotherapy every 4 weeks for up to 12 cycles after surgery unless disease is deemed unresectable, disease recurrence, or unacceptable toxicity
  The platinum-based chemotherapy will be based on tumour histology and Investigator discretion:
  * cisplatin with pemetrexed
  * carboplatin with pemetrexed
  * carboplatin with paclitaxel
  * cisplatin with gemcitabine (or carboplatin with gemcitabine for patients who have comorbidities or who are unable to tolerate cisplatin per the investigator's judgment)
  Interventions: Other: Placebo; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Gemcitabine; Procedure: Surgery

INTERVENTIONS:
Drug: Durvalumab — 1500mg on Day 1 of each 3-week cycle for 4 cycles during the neoadjuvant period and 1500mg on Day 1 of each 4-week cycle for 12 cycles during the adjuvant period
  Other Names: MEDI4736
  Arms: Arm 1: Durvalumab with platinum-based chemotherapy
Other: Placebo — Day 1 of each 3-week cycle for 4 cycles during the neoadjuvant period and Day 1 of each 4-week cycle for 12 cycles during the adjuvant period
  Arms: Arm 2: Placebo with platinum-based chemotherapy
Drug: Carboplatin — Area under the curve of 5/6 on Day 1 of each 3-week cycle for 4 cycles
Drug: Cisplatin — 75 mg/m2 on Day 1 of each 3-week cycle, for 4 cycles
Drug: Pemetrexed — 500 mg/m2 on Day 1 of each 3-week cycle for 4 cycles.
Drug: Paclitaxel — 200mg/m2 on Day 1 of each 3-week cycle for 4 cycles.
Drug: Gemcitabine — 1250 mg/m2 on Day 1 and Day 8 of each 3-week cycle, for 4 cycles.
Procedure: Surgery — Expected within 40 days from the last dose of Investigational Product following the completion of neoadjuvant treatment.

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled, multi-center international study assessing the activity of durvalumab and chemotherapy administered prior to surgery compared with placebo and chemotherapy administered prior to surgery in terms of pathological complete response.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Newly diagnosed and previously untreated patients with histologically or cytologically documented NSCLC with resectable (Stage IIA to select [ie, N2] Stage IIIB) disease
* World Health Organization (WHO)/ECOG PS of 0 or 1 at enrollment
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 Target Lesion (TL) at baseline
* No prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1, and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines
* Adequate organ and marrow function
* Confirmation of a patient's tumour PD-L1 status
* Provision of sufficient tumour biopsy sample for evaluation and confirmation of EGFR and ALK status
* Planned surgery must comprise lobectomy, sleeve resection, or bilobectomy

Exclusion Criteria:

* History of allogeneic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome)
* History of another primary malignancy
* History of active primary immunodeficiency
* Active infection including tuberculosis hepatitis B and C, or human immunodeficiency virus
* Deemed unresectable NSCLC by multidisciplinary evaluation
* Patients who have pre-operative radiotherapy treatment as part of their care plan
* Patients who have brain metastases or spinal cord compression
* Stage IIIB N3 and Stages IIIC, IVA, and IVB NSCLC
* Known allergy or hypersensitivity to any of the study drugs or excipients
* Existence of more than one primary tumour such as mixed small cell and NSCLC histology
* Patients whose planned surgery at enrollment includes any of the following procedures: pneumonectomy, segmentectomies, or wedge resections
* Patients with a documented test result confirming the presence of EGFRm or ALK translocation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2028-09-11 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) in modified intent-to-treat (mITT) population | Up to approximately 15 weeks after randomization
  Defined as the lack of any viable tumour cells after complete evaluation in the resected lung cancer specimen and all sampled regional lymph nodes.
Event-Free Survival (EFS) in modified intent to treat (mITT) population | Up to 5.5 years after first patient randomized.
  An event is defined as documented RECIST 1.1 local or distant recurrence of lung cancer; death due to any cause; disease progression that precludes surgery or discovered upon attempting surgery that prevents completion of surgery.

SECONDARY OUTCOMES:
Disease-free survival (DFS) in modified resected population | From date of randomization to approximately 5.5 years after date of resection
Major Pathological Response (mPR) in modified intent to treat (mITT) population | Up to approximately 15 weeks after randomization
Overall Survival (OS) in modified intent to treat (mITT) population | From date of randomization to 5.5 years after randomization
Event-free survival (EFS) in PD-L1-TC ≥1% patients in modified intent to treat (mITT) population | From date of randomization to 5.5 years after randomization
pCR in PD-L1-TC ≥1% patients in modified intent to treat (mITT) population | Up to approximately 15 weeks after randomization
Disease-Free Survival (DFS) in PD-L1-TC ≥1% patients in modified resected population | From date of randomization to 5.5 years after date of resection
Major Pathological Response (mPR) in PD-L1-TC ≥1% patients in modified intent to treat (mITT) population | Up to approximately 15 weeks after randomization
Overall Survival (OS) in PD-L1-TC ≥1% patients in modified intent to treat (mITT) population | From date of randomization to 5.5 years after randomization.
To assess disease-related symptoms and HRQoL (EORTC QLQ-C30) in patients treated with durvalumab + chemotherapy prior to surgery followed by durvalumab post-surgery compared with placebo + chemotherapy prior to surgery followed by placebo post-surgery | From date of screening to 6 months after last dose of IP
  To assess disease-related symptoms, functioning, and global health status/quality of life in patients.
To assess disease-related symptoms and HRQoL (EORTC QLQ-LC13) in patients treated with durvalumab + chemotherapy prior to surgery followed by durvalumab post-surgery compared with placebo + chemotherapy prior to surgery followed by placebo post-surgery | From date of screening to 6 months after last dose of IP
  To assess disease-related symptoms, functioning, and global health status/quality of life in patients.
To assess the PK of durvalumab in blood | From date of randomization to 2 months after resection
  To assess concentration of durvalumab in bloodstream.
Presence of ADA for durvalumab | From date of randomization to 3 months after last dose of IP
  To evaluate the presence of antibodies following treatment with study medications.

OTHER OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | From date of randomization to 3 months after last dose of IP

CONTACTS AND LOCATIONS:
Overall Officials: John Heymach, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (186):
- United States (28):
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, Aurora, Colorado
  - Research Site, Boca Raton, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Ashland, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Morristown, New Jersey
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, Durham, North Carolina
  - Research Site, Bend, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Kirkland, Washington
  - Research Site, Seattle, Washington
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Plata
  - Research Site, Pergamino
  - Research Site, Rosario
  - Research Site, San Salvador de Jujuy
  - Research Site, Viedma
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Rankweil
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Ghent
  - Research Site, Liège
  - Research Site, Mons
- Brazil (12):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Santa Maria
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Teresina
  - Research Site, Vitória
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Kitchener, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (22):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Xintai
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Research Site, San José, Costa Rica
- France (5):
  - Research Site, Avignon
  - Research Site, Lyon
  - Research Site, Nice
  - Research Site, Toulon
  - Research Site, Vantoux
- Germany (4):
  - Research Site, Bielefeld
  - Research Site, Cologne
  - Research Site, Frankfurt am Main
  - Research Site, Immenstadt im Allgäu
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- India (11):
  - Research Site, Ahmedabad
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, Manipal
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, Namakkal
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Thane
  - Research Site, Visakhapatnam
- Italy (9):
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Verona
- Japan (13):
  - Research Site, Habikino-shi
  - Research Site, Himeji-shi
  - Research Site, Hiroshima
  - Research Site, Iwakuni-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Kurashiki Shi
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osakasayama-shi
  - Research Site, Toyoake-shi
  - Research Site, Wakayama
- Mexico (6):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Pachuca
- Netherlands (2):
  - Research Site, Arnhem
  - Research Site, Nijmegen
- Peru (2):
  - Research Site, Bellavista
  - Research Site, Lima
- Philippines (4):
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Makati
  - Research Site, Quezon City
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Olsztyn
  - Research Site, Warsaw
- Research Site, Suceava, Romania
- Russia (9):
  - Research Site, Kazan'
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Obninsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Yaroslavl
- South Korea (5):
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (8):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Oviedo
  - Research Site, Pamplona
  - Research Site, Santiago de Compostela (A Coruña)
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Chiang Rai
  - Research Site, Khon Kaen
  - Research Site, Lampang
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information
URL: https://vivli.org/

REFERENCES:
- [Derived] Mitsudomi T, Heymach JV, Reck M, Taube JM, Gao S, Horio Y, You J, Li G, Van Luong D, Saeteng S, Tanaka F, Watzka SB, Urban L, Szalai Z, Akamatsu H, Kang JH, Orlandi FJ, Mukhametshina GZ, Pircher A, Teixeira CHA, Aperghis M, Doherty GJ, Doake R, Fouad TM, Harpole D. Surgical Outcomes With Neoadjuvant Durvalumab Plus Chemotherapy Followed by Adjuvant Durvalumab in Resectable NSCLC. J Thorac Oncol. 2025 Nov;20(11):1639-1654. doi: 10.1016/j.jtho.2025.06.015. Epub 2025 Jun 20. PMID 40545237
- [Derived] Heymach JV, Harpole D, Mitsudomi T, Taube JM, Galffy G, Hochmair M, Winder T, Zukov R, Garbaos G, Gao S, Kuroda H, Ostoros G, Tran TV, You J, Lee KY, Antonuzzo L, Papai-Szekely Z, Akamatsu H, Biswas B, Spira A, Crawford J, Le HT, Aperghis M, Doherty GJ, Mann H, Fouad TM, Reck M; AEGEAN Investigators. Perioperative Durvalumab for Resectable Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Nov 2;389(18):1672-1684. doi: 10.1056/NEJMoa2304875. Epub 2023 Oct 23. PMID 37870974